CLINICAL TRIAL: NCT07353970
Title: Mechanisms of Prognostic Regulation andPrecision Phenotype Ldentification in Severe Infections Driven by SpecializedPro-Resolving Mediators
Acronym: MPR-PPI-SPMs
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-03-135
Record Dates: First submitted 2026-01-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Severe Infection; Multiple Organ Dysfunction Syndrome; Critical Illness
Keywords: Specialized pro-resolving mediators; SPM; Resolvin D1; Immune resolution; Inflammation resolution; Critical care
MeSH Terms: conditions — Sepsis; Infections; Multiple Organ Failure; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Peripheral blood samples collected during routine clinical care will be used for the analysis of specialized pro-resolving mediators and related laboratory assessments. No samples will be used for DNA extraction or genetic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Infection ICU Cohort Adult patients: Adult patients with severe infection admitted to the intensive care unit (ICU). All participants receive standard clinical care as determined by their treating physicians. No experimental interventions are assigned.

SUMMARY:
This is a prospective observational study involving adult patients with severe infection who are admitted to the intensive care unit (ICU). Severe infection and sepsis are major causes of death worldwide. Many patients experience uncontrolled inflammation or immune suppression, but current tests are limited in identifying which patients are at highest risk.

This study focuses on specialized pro-resolving mediators (SPMs), a group of naturally occurring lipid molecules that help the body turn off inflammation and promote healing. Blood samples that are collected during routine clinical care will be used to measure levels of SPMs. No additional blood draws or experimental treatments will be performed.

The purpose of this study is to understand how SPM levels change over time in patients with severe infection and how these changes relate to organ function and outcomes such as survival. By combining SPM measurements with routine laboratory results, immune cell counts, and imaging findings, the study aims to identify different clinical phenotypes and to develop tools that may help doctors recognize high-risk patients earlier in the future.

All participants will receive standard medical care determined by their treating physicians. No experimental drugs or interventions are given as part of this study.

DETAILED DESCRIPTION:
Severe infection and sepsis remain leading causes of morbidity and mortality worldwide. Although antimicrobial therapy and organ support have improved, many critically ill patients continue to experience poor outcomes. Increasing evidence indicates that failure to appropriately resolve inflammation plays a key role in organ dysfunction and mortality. Specialized pro-resolving mediators (SPMs) are endogenous lipid mediators that actively terminate inflammation, promote clearance of pathogens and apoptotic cells, and support tissue repair. However, their role in human severe infection has not been systematically investigated in prospective clinical cohorts.

This study is a prospective observational cohort study enrolling adult patients with severe infection admitted to the intensive care unit (ICU). Approximately 300 patients are expected to be included. Peripheral blood samples obtained during routine clinical care on days 1, 3, and 7 after ICU admission will be analyzed. Plasma SPMs, including resolvins, protectins, and maresins, will be quantified using liquid chromatography-tandem mass spectrometry. Routine clinical data, including demographic characteristics, laboratory tests, immune cell subsets, coagulation indicators, severity scores (SOFA and APACHE II), organ support therapies, and 28-day outcomes will be recorded.

The study has four major objectives:

to describe the temporal profiles of SPMs in severe infection

to determine associations between SPM levels and adverse outcomes including 28-day mortality and organ failure

to identify biologically and clinically meaningful phenotypes driven by SPM signatures through multivariate clustering and machine-learning approaches

to explore mechanistic pathways linking SPMs with immune responses, coagulation disturbances, organ dysfunction, and clinical prognosis

No experimental medications or interventional procedures are administered as part of this study. All treatments are determined exclusively by the treating physicians according to routine clinical practice. No genetic testing or DNA extraction will be performed from collected samples.

The expected outcome of this study is the development of an SPM-based precision phenotyping framework that may support individualized risk assessment and potential future therapeutic strategies targeting impaired inflammation resolution.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to the intensive care unit (ICU)
* Diagnosis of severe infection or sepsis, as determined by the treating physician according to current clinical criteria
* Ability to obtain blood samples as part of routine clinical care within 24-48 hours after ICU admission
* Informed consent provided by the patient or legally authorized representative (when applicable)

Exclusion Criteria:

* Known pregnancy
* Known immunosuppressive disease (e.g., hematologic malignancy, advanced HIV infection)
* Use of long-term immunosuppressive therapy or systemic corticosteroids prior to ICU admission
* Pre-existing end-stage disease with expected survival < 28 days (e.g., end-stage cancer receiving palliative care)
* Enrollment in interventional clinical trials that may influence immune or inflammatory responses
* Refusal of informed consent by the patient or legal representative
* Patients in whom blood sampling or follow-up is not feasible (e.g., expected transfer, withdrawal of life-sustaining treatment within 24 hours)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients with severe infection or sepsis admitted to a tertiary academic medical center. Both male and female patients aged 18 years or older are eligible. All participants receive standard clinical care, and no experimental treatments are provided within this study.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-16 (Estimated); Study Completion 2028-01-16 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | From the date of ICU admission until death from any cause, assessed up to 28 days
  All-cause mortality assessed within 28 days after admission to the intensive care unit.

SECONDARY OUTCOMES:
ICU length of stay | From ICU admission to ICU discharge, assessed up to 28 days.
  Length of stay in the intensive care unit, measured in days from ICU admission to ICU discharge.
Organ dysfunction | Organ dysfunction assessed using routinely collected clinical data from ICU admission through day 28.
  Organ dysfunction assessed using routinely collected clinical data during the first 28 days after ICU admission
Secondary infection during ICU stay | From the date of ICU admission until the occurrence of a secondary infection or ICU discharge, whichever occurred first, assessed up to 28 days
  Secondary infection defined as a newly diagnosed infection occurring after ICU admission, confirmed by clinical signs, microbiological evidence, and/or initiation of targeted antimicrobial therapy, based on routinely collected clinical data.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves sensitive clinical information, and data sharing is not covered by the current ethics approval. Data will be used solely for the purposes specified in the approved study protocol.